CLINICAL TRIAL: NCT00789074
Title: Effects of an Extended Period of Varenicline Use Prior to Quitting Smoking on Post-quitting Urges to Smoke
Brief Title: Use of Varenicline for 4-weeks Prior to Quitting
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Principal Investigator, Professor Peter Hajek, Professor of Clinical Psychology, Queen Mary University of London
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: qmul120508
Record Dates: First submitted 2008-11-07; First posted 2008-11-11 (Estimated); Results first posted 2012-06-25 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-11

CONDITIONS: Tobacco Dependence; Smoking Cessation
Keywords: Smoking cessation; Tobacco dependence; Varenicline; Preloading
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Varenicline pre-treatmemt (Experimental): Participants will use varenicline (1mg BD) 4-weeks prior to quitting
  Interventions: Drug: Varenicline
- Placebo (Placebo Comparator): Participants will use 3 weeks of placebo, followed by 1 week of varenicline, prior to quitting
  Interventions: Drug: Varenicline; Drug: Placebo

INTERVENTIONS:
Drug: Varenicline — Varenicline 1mg twice daily
  Other Names: Champix
Drug: Placebo — Placebo 1mg BD
  Arms: Placebo

SUMMARY:
Varenicline (Champix) is a relatively new medicine that is effective in helping people to quit smoking. It is normally started 1-week before stopping smoking and used for up to 12-24 weeks. We are trying to find out if using varenicline for an extended time (4-weeks) before stopping smoking is better than the standard 1-week of use prior to stopping.

The study will recruit 100 smokers who want to stop. They will be randomly allocated to receive varenicline(4-weeks) or placebo (3-weeks followed by 1-week of active treatment as indicated by standard prescribing practice), followed by a 12-week open label treatment period where all participants will receive varenicline.

ELIGIBILITY:
Inclusion Criteria:

* Smokers seeking treatment
* Aged 18 and over
* Consenting to take part in the trial

Exclusion Criteria:

* Pregnant or breastfeeding
* End-stage renal disease
* Used varenicline in the past 6 months
* Unable to fill in questionnaires in English
* Current psychiatric illness
* Current serious illness including uncontrolled hypertension and recent cardiac event
* Sensitivity to varenicline currently enrolled in other research projects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2009-07; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Al-Rehan A A Dhanji, MB BS BSc MRCP, Principal Investigator — Queen Mary University of London
Locations (1):
- Tobacco Dependence Research and Treatment Unit, London, United Kingdom

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Hajek P, McRobbie HJ, Myers KE, Stapleton J, Dhanji AR. Use of varenicline for 4 weeks before quitting smoking: decrease in ad lib smoking and increase in smoking cessation rates. Arch Intern Med. 2011 Apr 25;171(8):770-7. doi: 10.1001/archinternmed.2011.138. PMID 21518946

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Varenicline Pre-treatmemt | Placebo
Started | 53 | 48
Completed | 42 | 35
Not Completed | 11 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline Pre-treatmemt | Placebo | Total
Number analyzed (Participants) | 53 | 48 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 47 | 96
  >=65 years | 4 | 1 | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 45.91 (11.439) | 45.29 (10.941) | 45.61 (11.153)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 36
  Male | 34 | 31 | 65
Region of Enrollment [Number; unit: participants]
  United Kingdom | 53 | 48 | 101

OUTCOME MEASURES:

1. Primary Outcome: Rating of Urges to Smoke 24 Hours and One Week After the Target Quit Date Assessed by Mood and Physical Symptoms Scale
Description: The scale measures tobacco withdrawal symptoms (depressed, irritable, restless, hungry, poor concentration, slept worse than usual) on 5-point scales from Not at all (rated as 1) to Extremely (rated as 5). It also asks 'How much of the time have you felt the urge to smoke in the last week? and 'How strong have these urges been?'; both rated on 6-point scales with higher numbers=higher craving.
Time Frame: 24 hours and 7 days after quit date (week 4)
Population: Were abstinent and provided data at 24 hours post quit date
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 34 | 29
units on a scale | 2.47 (1.13) | 2.88 (1.15)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Test type: Superiority or Other; p = 0.14, ANOVA

2. Secondary Outcome: Change in Pre-quit End-expired Carbon Monoxide Reading (CO)
Description: Carbon monoxide concentration is measured in particles per million. It indicates smoke intake.
  CO was measured at each contact to monitor changes in smoke intake and differences between the study arms.
Time Frame: Baseline - week 8
Population: Participants that provided data at all time points
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 47 | 40
ppm | -14.85 (11.08) | -7.68 (10.34)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA; Changes were compared using repeated measures analysis of variance

3. Secondary Outcome: Change in Pre-quit Cotinine Levels
Description: Differences in baseline cotinine levels were compared with cotinine levels measured 4 weeks after taking the first medication dose.
Time Frame: Weeks 1-4 (the first 4-weeks after first medication dose)
Population: All participants that provided data at all time points
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Varenicline Pre-treatmemt | Placebo
Number analyzed (Participants) | 47 | 41
ng/ml | -184.69 (156.02) | -44.73 (114.56)
Statistical Analysis 1: Comparison: Varenicline Pre-treatmemt vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA — F=16.60; Changes were compared using repeated measures analysis of variance

4. Secondary Outcome: Change in Pre-quit Ratings of Cigarette Satisfaction
Description: Satisfaction measured on a scale of 1-5; "Have you found your cigarettes more or less enjoyable than usual in the last week?" 1= much more and 5 = much less
Time Frame: Baseline - week 4
Population: Participants who provided ratings of cigarette satisfaction at each visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Varenicline Pre-treatmemt | Placebo
Number analyzed (Participants) | 40 | 38
units on a scale | -1.48 (1.66) | -0.842 (1.26)
Statistical Analysis 1: Comparison: Varenicline Pre-treatmemt vs Placebo; Test type: Superiority or Other; p < 0.04, ANOVA — F=2.92; Changes were compared using repeated measures analysis of variance

5. Secondary Outcome: Change in Pre-quit Cigarette Consumption
Description: Participants reported average number of cigarettes smoked per day every week throughout the four week pre-quit period.
Time Frame: Baseline - week 4
Population: All participants that provided data at each session
Measure: Mean (Standard Deviation); unit: Cigarettes consumed per day
Arm/Group | Varenicline Pre-treatment | Placebo
Number analyzed (Participants) | 46 | 40
Cigarettes consumed per day | -9.78 (9.67) | -5.68 (7.29)
Statistical Analysis 1: Comparison: Varenicline Pre-treatment vs Placebo; Test type: Superiority or Other; p = 0.02, ANOVA; Changes were compared using repeated measures analysis of variance

6. Secondary Outcome: Change in MPSS Scores of Urges to Smoke and Cigarette Withdrawal Symptoms Throughout the First Four Weeks of Abstinence
Description: Change in the Mood and Physical Symptoms Scale (MPSS)*, scores of urges to smoke and cigarette withdrawal symptoms throughout the first four weeks of abstinence (measured weekly from weeks 4-8).
  * The MPSS measures cigarette withdrawal symptoms. The scale is 1-5, 1 being not at all and 5 being extremely (depressed, irritable, restless, hungry, poor concentration, slept worse than usual).
Time Frame: Week 4 - 8
Population: Participants who were abstinent at 1 week and provided data on withdrawal symptoms
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Varenicline Pre-treatment | Placebo
Number analyzed (Participants) | 35 | 25
Scores on a scale | 0.15 (0.68) | 0.15 (0.53)
Statistical Analysis 1: Comparison: Varenicline Pre-treatment vs Placebo; Test type: Superiority or Other; p = 0.97, ANOVA; Changes were compared using repeated measures analysis of variance

ADVERSE EVENTS:
Arm/Group | Varenicline Pre-treatmemt | Placebo
Serious Adverse Events (participants affected / at risk) | 1/53 | 1/48
Other Adverse Events (participants affected / at risk) | 34/53 | 22/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline Pre-treatmemt (N=53) | Placebo (N=48)
Acute Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline Pre-treatmemt (N=53) | Placebo (N=48)
Nausea (Gastrointestinal disorders) | 34 (34) | 22 (22)
Abnormal dreams (Psychiatric disorders) | 14 (14) | 7 (7)
Headache (General disorders) | 12 (12) | 7 (7)
Sleep disturbance (Psychiatric disorders) | 10 (10) | 6 (6)
Constipation (Gastrointestinal disorders) | 7 (7) | 1 (1)
Drowsiness (General disorders) | 6 (6) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 6 (6) | 7 (7)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 4 (4)
Sweating (General disorders) | 5 (5) | 0 (0)
Depression (Psychiatric disorders) | 4 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 2 (2)
Fatigue (Nervous system disorders) | 4 (4) | 3 (3)
Light headedness (Nervous system disorders) | 4 (4) | 0 (0)
Muscularskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Flu like symptoms (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 3 (3) | 1 (1)
Poor concentration (General disorders) | 3 (3) | 1 (1)
Skin irritation/rash (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2)
Bleeding gums (General disorders) | 1 (1) | 3 (3)
Chest pain - not specified (General disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes